CLINICAL TRIAL: NCT04451889
Title: Probe-based Confocal Laser Endomicroscopy in Critically Ill COVID-19 Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal Research Clinical Center of Federal Medical & Biological Agency, Russia (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: COVID-pCLE
Record Dates: First submitted 2020-06-29; First posted 2020-06-30 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2020-06

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Confocal laser endomicroscopy diagnostic study (Experimental): Cohort 1: COVID-19 patients. Cohort 2: patients with lung diseases unrelated to COVID-19.
  All the patients will be examined using confocal laser endomicroscopy during bronchoscopy with a special Alveoflex miniprobe during the hospitalisation period. Records will be done and analysed prospectively with the included software for the endomicroscopic system.
  Using Alveoflex is a minimally invasive intervention.
  Interventions: Device: miniprobe Alveoflex

INTERVENTIONS:
Device: miniprobe Alveoflex — Alveoflex uses 488nm laser, generating real time moving images with an optical area of 600μm at a video frame rate of 12 images per second and a focus depth of 50μm
  Other Names: Cellvizio system (Mauna Kea Technologies, Paris, France)

SUMMARY:
The study is devoted to the comparative analysis of the data received in patients with COVID-19 lung pathology using the method of probe-based confocal laser endomicroscopy of distal airways and two reference methods: high resolution computed tomography and morphology (in some patients).

ELIGIBILITY:
Inclusion Criteria:

* Patient Informed Consent;
* the diagnosis of COVID-19 or one of the following lung diseases: chronic obstructive pulmonary disease, pneumonia, solitary nodule, pulmonary sarcoidosis, idiopathic interstitial pneumonia, hypersensitivity pneumonitis, pulmonary vasculitis, pulmonary eosinophilia, hemochromatosis, histiocytosis X, pulmonary lymphangioleiomyomatosis; alveolar proteinosis, other rare lung disease
* high resolution computed tomography scans performed not later than one month before pCLE (for non-COVID-19);
* planned or performed histology (for non-COVID-19)
* Severe respiratory failure,

Exclusion Criteria:

* pregnancy or breast feeding,
* lung bleeding,
* any acute or chronic disease that may be a contraindication to bronchoscopy,
* any diseases of hematopoietic system,
* taking part in other clinical trials

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Number of COVID-19 Participants With Notable Differences in the pCLE images in comparison with the pCLE images of non-COVID-19 Participants | up to one year
  pCLE images are assessed morphometrically. Such criteria as quantity of alveolar macrophages, quantity of floating intraalveolar substances etc. are measured using a 6-point score, where zero means the absence of the symptom and 5 means the maximal expressiveness. Thickness of interalveolar septum, diameter of microvessels and thickness of elastic fibers are measured using a special tool with the included software for the endomicroscopic system. Radiologic signs e.g. low-density areas and consolidation areas are assessed in Hounsfield Units. Other radiologic signs e.g. groundglass opacity, crazy paving patterns etc. are measured by a 5-point scale, where zero means the absence of the symptom and 4 means the maximal expressiveness. The morphological analysis of the lung tissue specimens (received as a result of autopsy/transbronchial biopsy) is made according to the structures in pCLE images for 20 fields of view.

SECONDARY OUTCOMES:
Number of Participants With the Correspondence of pCLE Images to High Resolution Computer Tomography and Morphologic Data as a Measure of Specificity and Sensitivity of the Method | up to one year
  pCLE images are assessed morphometrically. Such criteria as quantity of alveolar macrophages, quantity of floating intraalveolar substances etc. are measured using a 6-point score, where zero means the absence of the symptom and 5 means the maximal expressiveness. Thickness of interalveolar septum, diameter of microvessels and thickness of elastic fibers are measured using a special tool with the included software for the endomicroscopic system. Radiologic signs e.g. low-density areas and consolidation areas are assessed in Hounsfield Units. Other radiologic signs e.g. groundglass opacity, crazy paving patterns etc. are measured by a 5-point scale, where zero means the absence of the symptom and 4 means the maximal expressiveness. The morphological analysis of the lung tissue specimens (received as a result of autopsy/transbronchial biopsy) is made according to the structures in pCLE images for 20 fields of view.

CONTACTS AND LOCATIONS:
Overall Officials: Olesya Danilevskaya, MD, PhD, Principal Investigator — Federal Research Clinical Center FMBA Russia
Locations (1):
- Federal Research Clinical Center FMBA Russia, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No
There is no current plan to share individual participant data (IPD).